CLINICAL TRIAL: NCT04451798
Title: JENA Mechanical Assist Circulatory Support Trial-JENAMACS-hemodynamic
Brief Title: Acute Impact of the Impella CP Assist Device in Pts. With Cardiogenic Shock on the Patients Hemodynamic
Acronym: JenaMACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Collaborators: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, Principal Investigator, Clinical Professor, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMW 07
Record Dates: First submitted 2020-03-01; First posted 2020-06-30 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Cardiogenic Shock
Keywords: Impella
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Impella implantation and hemodynamic measurement
  Interventions: Device: Impella CP microaxial pump

INTERVENTIONS:
Device: Impella CP microaxial pump — ramp test

SUMMARY:
Prospective, monocentric open-label observational study for the assessment of acute hemodynamic effects following implantation of the IMPELLA CP cardiac support device

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock following acute MI or acute heart failure with

  * systolic BP < 90 mm Hg over > 30 min or inotropes for support of cardiac output and BP with
  * signs of left heart failure and pulmonary congestion
  * and end-organ hypo perfusion with somnolence or cold, pale skin, or oliguria or serum lactate >2 mmol/l

Exclusion Criteria:

Ages: 16 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Parameters due to PA catheterisation | Day 1
  Pulmonary capillary Wedge pressure in dependence of Impella pump level
Echocardiographic Parameters of left and right heart function | Day 1
  LV- size in dependence of Impella pump level

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, MD, Principal Investigator — Universityhospital Jena
Locations (1):
- University of Jena, Jena, Germany

IPD SHARING:
Plan to Share IPD: No